CLINICAL TRIAL: NCT06660719
Title: A Multi-Center, Randomized, Double-Blind, Parallel, Placebo-Controlled, Phase III Clinical Study to Evaluate Efficacy and Safety of SP-8203 (Otaplimastat) in Patients With Acute Ischemic Stroke Requiring Thrombolytic Therapy as Standard of Care
Brief Title: Efficacy and Safety of SP-8203 (Otaplimastat) in Patients With Acute Ischemic Stroke Receiving Thrombolytic Standard of Care
Acronym: SP-8203-3001
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-8203-3001
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Ischemic Stroke
Keywords: SP-8203 (Otaplimastat); rtPA (recombinant tissue Plasminogen Activator); Thrombolytic therapy
MeSH Terms: conditions — Ischemic Stroke | interventions — otaplimastat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SP-8203 (Experimental): SP-8203 80 mg (40 mg/dose twice a day for three days)
  Interventions: Drug: SP-8203
- Placebo (Placebo Comparator): Placebo group: twice a day for three days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SP-8203 — SP-8203 80 mg will be intravenously administered as 40 mg/dose twice daily (intervals of 12 hours)
  Other Names: Otaplimastat (SP-8203)
  Arms: SP-8203
Drug: Placebo — Placebo will be intravenously administered twice daily (intervals of 12 hours)
  Arms: Placebo

SUMMARY:
This clinical study is designed to evaluate the efficacy and safety of the combination therapy of SP-8203 (otaplimastat) and thrombolytic standard of care in acute ischemic stroke patient.

As a standard of care, thrombolytic therapy (for instance, recombinant tissue plasminogen activator) will be administered. When reperfusion is not achieved in spite of thrombolytic therapy, endovascular therapy can be performed.

DETAILED DESCRIPTION:
Intravenous administration of SP-8203 (otaplimastat), a multipotent neuroprotectant inhibiting matrix metalloprotease activity, significantly reduced infarct volume and recombinant tissue plasminogen activator (rtPA)/ ischemic-induced damage in animal models.

This clinical study is designed to evaluate the efficacy and safety of the combination therapy of SP-8203 (otaplimastat) and thrombolytic standard of care in acute ischemic stroke patient.

As a standard of care, thrombolytic therapy (for instance, recombinant tissue plasminogen activator) will be administered. When reperfusion is not achieved in spite of thrombolytic therapy, endovascular therapy can be performed.

A total of 852 participants will be enrolled in double-blind, randomized and parallel design with 426 participants assigned to 80 mg/day SP-8203 arm or placebo arm, respectively.

Eligible participants are the patients with neurologic deficit of ≥8 point on National Institute of Health Stroke Scale (NIHSS) score. The participant will receive the study intervention a total of 6 times, with 12 hours intervals. Imaging test will be performed using validated machine and method. The participant will have initial brain Magnetic Resonance Imaging (MRI) and Magnetic Resonance Angiography (MRA) performed within 6 hours before or after the administration of study intervention, and brain Computed Tomography (CT) will be performed at 24±3 hours after completion of the first administration of study intervention.

Brain Magnetic Resonance Imaging (MRI) and Magnetic Resonance Angiography (MRA) will be followed-up on Day 5, and additionally the participant will undergo additional functional and neurological evaluations for up to 90 days.

When unexpected serious adverse reaction occurs during the clinical study, Data Safety Monitoring Board (DSMB) will be convened to validation safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurologic deficit of ≥ 8 points by National Institute of Health Stroke Scale (NIHSS) score
* Patients with pre-stroke modified Rankin Scale (mRS) must be 0 or 1, which means they were able to carry out all usual duties and activities
* Adults aged ≥19 years and ≤85 years
* Patients who can receive thrombolytic standard of care within 4.5 hours after the onset of early symptoms of acute ischemic stroke
* Patients available for brain Magnetic Resonance Imaging (MRI) scanning
* Patients who consent to participate in this study

Exclusion Criteria:

* Patients with systemic allergic diseases or hypersensitivity to specific drugs.
* Patients who were diagnosed with myocardial infarction (MI) within the last 6 months.
* Patients who had arrhythmia causing clinical symptoms such as dyspnea or palpitation within the last 6 months.
* Patients showing the following abnormal ECG findings in stable condition at Emergency Room:

  * The range of pulse rate - under 55/min or exceed 120/min
  * 2nd or 3rd degree Atrioventricular (AV) block indicated in ECG
  * Congenital or acquired QT syndrome indicated in ECG
  * Pre-excitation syndrome indicated in ECG
* Patients with severe heart failure of New York Heart Association (NYHA) Class III or Class IV.
* Patients with fever (≥ 38℃) or infection signs which require antibiotic therapy at screening.
* Patients with pulmonary diseases (asthma, Chronic Obstruction Pulmonary disease, and active tuberculosis etc.) who have being recently been treated more than 1 month at screening.
* Patients with decreased hemoglobin (Hb< 10g/dL), decreased platelet count (PLT< 100,000/mm3) or hematocrit of <25% in complete blood count.
* Patients who have undergone hemodialysis and/or treatments due to nephropathies, acute or chronic renal failure at screening.
* Patients with a cancer in following conditions: diagnosed within 6 months before the screening time, or any treatment for cancer within the previous 6 months, or with recurrent/ metastatic cancer.
* Pregnant and lactating women. However, Women of Childbearing Potential (WOCBP) can participate in the study only when non-pregnancy is confirmed. Women of Childbearing Potential (WOCBP) is defined as woman who is not definitely menopause and did not receive a surgical contraception.
* Patients who do not consent to use double barrier contraception until 90 days from the first study intervention administration.
* Patients who have participated in other clinical trials of other drugs within the past 3 months. However, if they participated in observational studies and did not take drugs, they can participate in this trial.
* Patients who cannot participate in the study at the discretion of investigators
* Patients who are unable to receive thrombolytic standard of care, rtPA

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 852 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with modified Rankin Scale (mRS) 0-1 | Day 90
  Proportion of participants with modified Rankin Scale (mRS) 0-1 at Day 90 in patients with acute ischemic stroke requiring thrombolytic standard of care

SECONDARY OUTCOMES:
Incidence of parenchymal hematoma observed on brain Computed Tomography (CT) scan | Day 1
  Incidence of parenchymal hematoma observed on brain Computed Tomography (CT) scan performed at 24±3 hours in accordance with European Cooperative Acute Stroke Study (ECASS) I and II criteria, after the administration of SP-8203 in conjunction with thrombolytic standard of care
Proportion of participants with modified Rankin Scale (mRS) 0-1 | Day 30
  Proportion of participants with modified Rankin Scale (mRS) 0-1 at Day 30 in patients with acute ischemic stroke requiring thrombolytic standard of care
Proportion of participants with modified Rankin Scale (mRS) 0-2 | Day 30 and Day 90
  Proportion of participants with modified Rankin Scale (mRS) 0-2 at Day 30 and Day 90 in the patients with acute ischemic stroke requiring thrombolytic standard of care
Change from Baseline in National Institute of Health Stroke Scale (NIHSS) scores | Day 0 (baseline), Day 3, Day 5, Day 30 and Day 90
  The change in the National Institute of Health Stroke Scale (NIHSS) scores until 90 day in subjects with acute ischemic stroke requiring rtPA standard of care. The maximum total score is 42 points, which indicates the most critical condition and the minimum total score is 0, which indicates no neurologic deficit.
Fold change in infarct growth classified by modified treatment in cerebral ischemia (mTICI) grade within 5 days | Day 5
  MRI (DWI) imaging outcomes
The incidence of serious adverse events | follow-up to 90 days after the first study intervention administration
  The incidence of serious adverse events
The rate of death | follow-up to 90 days after the first study intervention administration
  The rate of death due to any cause
The incidence rate of adverse events, and adverse drug reaction | follow-up to 90 days after the first study intervention administration
  The incidence rate of adverse events, and adverse drug reaction
The incidence of symptomatic Intracranial Hemorrhage (sICH) | within 5 days from the first study intervention administration
  The incidence of symptomatic Intracranial Hemorrhage (sICH) occurring within 5 days of administration according to the definition described on the protocol
The Incidence of major systemic bleeding | within 5 days after the first study intervention administration
  The Incidence of major systemic bleeding according to the International Society of Thrombosis and Hemostasis (ISTH) definition

CONTACTS AND LOCATIONS:
Overall Officials: Jong Sung Kim, MD, Phd, Study Chair — GangNeung Asan Medical Center; Beom Jun Kim, MD, Phd, Principal Investigator — Seoul Asan Medical Center
Locations (2):
- South Korea (2):
  - Dong-A University Hospital, Busan
  - Ulsan University Hospital, Ulsan